CLINICAL TRIAL: NCT01069458
Title: The Effect of a High Protein Diet Versus a Low Fat Diet on Body Weight and Composition, Total Energy Expenditure, Metabolic Risk Factors and Eating Behavior After Smoking Cessation
Brief Title: The Effect of a High Protein Diet Versus a Low Fat Diet on Body Weight After Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tor Ole Klemsdal, Chief Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1375
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Smoking; Overweight; Obesity
Keywords: Dietary intervention; Smoking cessation; Body weight
MeSH Terms: conditions — Smoking; Overweight; Obesity; Smoking Cessation; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The High Protein Diet Group (Experimental): The high protein diet (25% energy from protein, 55% energy from fat, 20% energy from carbohydrate) will be hypo-caloric and achieved by restricting the amount of sugar containing foods and drinks, reducing the intake of bread, rice, pasta, fruits and fruit-juices and increasing the intake of vegetables (instead of bread, rice, pasta and potatoes) and increasing the amounts of protein (from chicken, fish, and meat) and fat from oil and dressings for lunch and dinner and by choosing nuts and protein-rich yoghurts, egg, cheese, chicken wings, shellfish, fish and fish products as snacks.
  Interventions: Other: The high protein diet group and the low fat diet group
- The Low Fat Diet Group (Active Comparator): The low fat diet (30% energy from fat, 20% energy from protein, 50% energy percent from carbohydrate) will be hypo-caloric and achieved by choosing low-fat diary and meat products, restricting amounts of visible fat and fatty snacks and increasing intake of whole meal bread, muesli, brown rice, whole meal pasta in the main meals and by choosing yoghurt with muesli, oat porridge with milk, fruits and hard bread with jam and soft gout-cheese as snacks.
  Interventions: Other: The high protein diet group and the low fat diet group

INTERVENTIONS:
Other: The high protein diet group and the low fat diet group — The High Protein Diet Group was advised to have 25 energy percent from protein, 55 energy percent from fat, 20 energy percent from carbohydrate in the diet and the Low Fat Diet Group was advised to have 30 energy percent from fat, 20 energy percent from protein, 50 energy percent from carbohydrate in the diet.
  Other Names: The high protein diet group; The low fat diet group

SUMMARY:
The purpose of this study is to determine whether subjects following a high protein diet will gain less in weight after smoking cessation compared to subjects following a low fat diet due to the effects of protein on metabolic rate and hunger.

DETAILED DESCRIPTION:
Sustained smoking cessation is one of the most effective therapies to avoid premature morbidity and mortality. However, weight gain associated with nicotine withdrawal may attenuate some of the beneficial health effects and is cited as a major obstacle to quit smoking. The mechanism for the weight gain is not elucidated but reduced resting metabolic rate, reduced total energy expenditure, increased caloric intake and changes in fat metabolism may be involved. Elucidating effective strategies to prevent or reduce post-cessation weight gain may improve health outcomes of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 10 cigarettes per day, BMI 25-40

Exclusion Criteria:

* Recent change in weight, contra-indications to use varenicline, a medication to assist smoking cessation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Body weight and waist circumference | 4 weeks, 3 months and 6 months after smoking cessation

SECONDARY OUTCOMES:
Resting metabolic rate, total energy expenditure, body composition, components of metabolic syndrome, eating behavior | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serena Tonstad, Professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Department of Preventive Cardiology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heggen E, Svendsen M, Tonstad S. Smoking cessation improves cardiometabolic risk in overweight and obese subjects treated with varenicline and dietary counseling. Nutr Metab Cardiovasc Dis. 2017 Apr;27(4):335-341. doi: 10.1016/j.numecd.2016.12.011. Epub 2017 Jan 4. PMID 28216282